CLINICAL TRIAL: NCT01859260
Title: Using CPAP to Prevent Acute Kidney Injury in Hospitalized Patients With Chronic Kidney Disease
Brief Title: Using Continuous Positive Airway Pressure to Reduce the Incidence of Acute Kidney Injury in Hospitalized Patients With Chronic Kidney Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TGHCPAPCKD
Record Dates: First submitted 2013-05-15; First posted 2013-05-21 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2013-05

CONDITIONS: Chronic Kidney Disease; Obstructive Sleep Apnea
Keywords: chronic kidney disease, acute kidney injury, obstructive sleep apnea
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sleep Apnea, Obstructive; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental): CPAP/autopap
  Interventions: Device: CPAP/autopap

INTERVENTIONS:
Device: CPAP/autopap
  Arms: Intervention

SUMMARY:
Obstructive sleep apnea (OSA) is a common and undertreated condition in patients with chronic kidney disease (CKD). Both physiologic and empiric data suggest that renal hypoxia due to OSA is associated with worsening kidney function. Hospitalized patients are often exposed to multiple nephrotoxins such as antibiotics, contrast agents, and diuretics, which place them at risk for acute worsening of kidney function. This study aims to determine whether immediate diagnosis and treatment of OSA in CKD patients will decrease the incidence of acute kidney injury during hospitalization. The investigators will evaluate the extent to which this effect can be attributed to a decrease in nocturnal hypoxia and improved blood pressure control. Secondary endpoints include hospital length of stay, and a composite outcome comprised of hemodialysis initiation, major cardiovascular events, and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. CKD defined by National Kidney Foundation Staging system: eGFR < 60
2. Overnight sleep study consistent with OSA

Exclusion Criteria:

1. Currently treated with positive airway pressure for sleep-disordered breathing
2. Hemodynamically unstable, defined as SBP < 90, or use of vasopressors
3. Intubated or mechanically ventilated
4. Respiratory insufficiency, defined as P/F ratio < 250, or requiring mechanical ventilation
5. End stage renal disease on renal replacement therapy
6. Contraindication to CPAP, including active emesis, recent intracranial surgery, altered level of consciousness

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05-30 (Actual); Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury | participants will be followed for the duration of hospital stay, an expected average of 5 days
  incidence of acute kidney injury during hospitalization (defined as an increase in creatinine by 0.5 mg/dl or more)

SECONDARY OUTCOMES:
Nocturnal hypoxia | participants will be followed for the duration of hospital stay, an expected average of 5 days
  Nocturnal hypoxia, defined as oxygen saturation < 88%
Blood pressure control | participants will be followed for the duration of hospital stay, an expected average of 5 days
  Blood pressure control, defined as incidence of SBP > 160
Hospital length of stay | participants will be followed for the duration of hospital stay, an expected average of 5 days
  Hospital length of stay
composite outcome | participants will be followed for the duration of hospital stay, an expected average of 5 days
  Composite outcome of a) Incidence of major cardiovascular event (acute coronary syndrome, major arrhythmia, or exacerbation of CHF), b) Initiation of hemodialysis c)In-hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Tampa general hospital, Tampa, Florida, United States

REFERENCES:
- [Background] Kanbay A, Buyukoglan H, Ozdogan N, Kaya E, Oymak FS, Gulmez I, Demir R, Kokturk O, Covic A. Obstructive sleep apnea syndrome is related to the progression of chronic kidney disease. Int Urol Nephrol. 2012 Apr;44(2):535-9. doi: 10.1007/s11255-011-9927-8. Epub 2011 Mar 3. PMID 21369754
- [Background] Zoccali C, Mallamaci F, Tripepi G. Sleep apnea in renal patients. J Am Soc Nephrol. 2001 Dec;12(12):2854-2859. doi: 10.1681/ASN.V12122854. No abstract available. PMID 11729258
- [Background] Fletcher EC. Obstructive sleep apnea and the kidney. J Am Soc Nephrol. 1993 Nov;4(5):1111-21. doi: 10.1681/ASN.V451111. PMID 8305638
- [Background] Fine LG, Norman JT. Chronic hypoxia as a mechanism of progression of chronic kidney diseases: from hypothesis to novel therapeutics. Kidney Int. 2008 Oct;74(7):867-72. doi: 10.1038/ki.2008.350. Epub 2008 Jul 16. PMID 18633339
- [Background] Nicholl DDM, Ahmed SB, Loewen AHS, Hemmelgarn BR, Sola DY, Beecroft JM, Turin TC, Hanly PJ. Declining kidney function increases the prevalence of sleep apnea and nocturnal hypoxia. Chest. 2012 Jun;141(6):1422-1430. doi: 10.1378/chest.11-1809. Epub 2012 Jan 5. PMID 22222188